CLINICAL TRIAL: NCT07277491
Title: Assessment of Nutritional Status in Rheumatic Diseases and Association to Disease Activity
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Mahmoud Lotfy, Rheumatology Specialist, Cairo University
Other Study IDs: MD-66-2023
Record Dates: First submitted 2025-09-05; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Spondyloarthritis (SpA); Psoriatic Arthritis (PsA); Systemic Lupus Erythematous (SLE); Systemic Sclerosis (SSc); Rheumatoid Arthritis (RA
Keywords: nutritional status; rheumatic diseases; disease activity
MeSH Terms: conditions — Spondylarthritis; Arthritis, Psoriatic; Scleroderma, Systemic; Arthritis, Rheumatoid; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases with different rheumatic diseases: 135 patients with different rheumatic diseases who attended the outpatient Rheumatology Clinic, Cairo University Hospitals as well as the Health Insurance Hospital, Aswan Governorate Patients diagnosed with rheumatic diseases including RA,SpA,SLE and SSc were included
- control cases matched for age and sex: control cases selected from healthy volunteers matched for age and sex

SUMMARY:
The aim of the present work is to assess the nutritional status among different rheumatic diseases patients and to study its association with the corresponding diseases activity.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is an autoimmune, progressive, systemic disease of connective tissue. It is characterized by arthritis (symmetrical in most cases), extra-articular and systemic change. Spondyloarthritis (SpA) is an interconnected group of rheumatic disorders including ankylosing spondylitis (AS) and psoriatic arthritis (PsA), characterized by common clinical symptoms and a similar genetic background .Systemic Lupus Erythematous (SLE) is a chronic connective tissue disease characterized by a multi-system inflammatory disorder with immune system imbalance .Systemic sclerosis (SSc) is an immune-mediated rheumatic disease characterized by fibrosis of the skin and internal organs as well as vasculopathy .

Nutritional status has been widely related to immunity; under-nutrition is associated with immunosuppression and increased susceptibility to infection whereas over-nutrition is associated with low-grade chronic inflammation increasing the risk and affecting the prognosis in metabolic, cardiovascular, and autoimmune diseases .

Patients with rheumatic diseases are prone to develop malnutrition as their medications often affect appetite, nutrient absorption and digestion.Despite the high incidence of malnutrition and its consequences, there is no universally accepted definition for diagnosing nutritional deficiencies, and nutritional assessment still relies on analyses of a combination of several anthropometric, biochemical, immunological, functional and body composition data, in addition to dietary intake and the evaluation of clinical status.

Four malnutrition diagnostic tools are currently used in adults: Subjective Global Assessment (SGA) ; Mini Nutritional Assessment (MNA) ; Academy of Nutrition and Dietetics/American Society for Parenteral and Enteral Nutrition malnutrition consensus characteristics; and Global Leadership Initiative on Malnutrition criteria.

Certain objective nutritional assessment indices reflect the immune nutritional status of patients, such as the prognostic nutritional index (PNI) ; and the nutritional risk index (NRI) which are calculated using serum albumin level and lymphocyte count, were found to be related to the nutritional status and disease activity in SLE patients .

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with rheumatic diseases including RA, SpA, SLE and SSc.

Exclusion Criteria:

1. Patients who are unable to comply with the physician assessment.
2. Patients with other connective tissue diseases, neurological diseases, malignancy, heart failure or severe renal dysfunction was excluded, as these diseases affect the muscle mass causing sarcopenia.
3. Advanced liver diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population of study: Patients of both genders were recruited in this study. Study subjects were patients with different rheumatic diseases attending the outpatient Rheumatology Clinic. Patients who visited the clinic from January 2023 to December 2025 were asked to participate after being provided with an explanation of the work.
  Study location: Study was conducted in the outpatient clinics of the Rheumatology Department, Cairo University Hospitals as well as in the Health Insurance Hospital, Aswan Governorate.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Nutritional Status as Assessed by the Prognostic Nutritional Index (PNI) | Assessed during routine clinic visits between January 1, 2023, and December 30, 2025.
  The Prognostic Nutritional Index (PNI) is an index score calculated using the formula: Serum Albumin (g/L) + 5 × Total Lymphocyte Count (/mm³).
  Unit of Measure: Calculated Index Score Interpretation: Higher scores indicate better nutritional status
Nutritional Risk as Assessed by the Nutritional Risk Index (NRI) | Assessed during routine clinic visits between January 1, 2023, and December 30, 2025.
  The Nutritional Risk Index (NRI) is an index score calculated based on serum albumin levels and the percentage of weight loss.
  Unit of Measure: Calculated Index Score Interpretation: Higher scores indicate a lower nutritional risk
Nutritional Status as Assessed by the Subjective Global Assessment (SGA) | Assessed during routine clinic visits between January 1, 2023, and December 30, 2025.
  The Subjective Global Assessment (SGA) is a clinical tool that results in a score based on a patient questionnaire and physical examination.
  Unit of Measure: Score on a 7-point scale Interpretation: Higher scores indicate better nutritional status.
Nutritional Status as Assessed by the Mini Nutritional Assessment - Short Form (MNA-SF) | Assessed during routine clinic visits between January 1, 2023, and December 30, 2025
  The Mini Nutritional Assessment - Short Form (MNA-SF) is a screening tool consisting of a questionnaire administered to the patient.
  Unit of Measure: Score on a 14-point scale Interpretation: Scores are categorized as: 12-14 (normal nutritional status), 8-11 (at risk of malnutrition), or 0-7 (malnourished).

SECONDARY OUTCOMES:
corrolation between Body Mass Index (BMI) and disease activity | Assessed during routine clinic visits between January 1, 2023, and December 30, 2025
  Body Mass Index (BMI) will be calculated as weight in kilograms divided by the square of height in meters (kg/m^2). This will be reported as a continuous variable. Additionally, the percentage of participants in each standard BMI category (e.g., underweight, normal, overweight, obese) will be determined.
  * Unit of Measure: kg/m^2 and Percentage of participants.
corrolation between Prognostic Nutritional Index (PNI) and disease activity | Assessed during routine clinic visits between January 1, 2023, and December 30, 2025.
  PrognostiThe Prognostic Nutritional Index (PNI) score will be calculated using the formula: Serum Albumin (g/L) + 5 × Total Lymphocyte Count (/mm³). The resulting score, where higher values indicate better nutritional status, will be reported as a continuous variable.
  * Unit of Measure: Calculated Index Score.
corrolation between Nutritional Risk Index (NRI) and disease activity | Assessed during routine clinic visits between January 1, 2023, and December 30, 2025.
  The Nutritional Risk Index (NRI) score will be calculated based on serum albumin levels and patient weight changes. The resulting score, where higher values indicate lower nutritional risk, will be reported as a continuous variable.
  * Unit of Measure: Calculated Index Score
Corrolation between Nutritional Status Categorization by Subjective Global Assessment (SGA) and disease activity | Assessed during routine clinic visits between January 1, 2023, and December 30, 2025.
  The Subjective Global Assessment (SGA) will be used to classify participants into distinct nutritional categories: well-nourished, mildly/moderately malnourished, or severely malnourished.
  * Unit of Measure: Percentage of participants in each category.
Duration of Rheumatic Disease | Assessed during routine clinic visits between January 1, 2023, and December 30, 2025.
  The duration of a patient's rheumatic disease is recorded from the date of initial diagnosis as documented in their medical history. This variable will be used to assess the correlation between disease duration and various measures of nutritional status.
  Unit of Measure: Years

CONTACTS AND LOCATIONS:
Overall Officials: Dina Ossama Abdulazim, assistant professor, Principal Investigator — Rheumatology and Rehabilitation Department, Faculty of Medicine, Cairo University
Locations (1):
- Department: Rheumatology and Rehabilitation Department, Faculty of Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu H, Jiao J, Zhu M, Wen X, Jin J, Wang H, Lv D, Zhao S, Sun X, Wu X, Xu T. Nutritional Status According to the Short-Form Mini Nutritional Assessment (MNA-SF) and Clinical Characteristics as Predictors of Length of Stay, Mortality, and Readmissions Among Older Inpatients in China: A National Study. Front Nutr. 2022 Jan 25;9:815578. doi: 10.3389/fnut.2022.815578. eCollection 2022. PMID 35145987
- [Background] Olsen MN, Tangvik RJ, Halse AK. Evaluation of Nutritional Status and Methods to Identify Nutritional Risk in Rheumatoid Arthritis and Spondyloarthritis. Nutrients. 2020 Nov 21;12(11):3571. doi: 10.3390/nu12113571. PMID 33233336
- [Background] Malone A, Mogensen KM. Key approaches to diagnosing malnutrition in adults. Nutr Clin Pract. 2022 Feb;37(1):23-34. doi: 10.1002/ncp.10810. Epub 2021 Dec 22. PMID 34936131
- [Background] Klak A, Borowicz J, Manczak M, Grygielska J, Samel-Kowalik P, Raciborski F. Current nutritional status of patients with rheumatic diseases in the population of Poland. Reumatologia. 2015;53(1):26-33. doi: 10.5114/reum.2015.50554. Epub 2015 Apr 10. PMID 27407222
- [Background] Vellas B, Guigoz Y, Garry PJ, Nourhashemi F, Bennahum D, Lauque S, Albarede JL. The Mini Nutritional Assessment (MNA) and its use in grading the nutritional state of elderly patients. Nutrition. 1999 Feb;15(2):116-22. doi: 10.1016/s0899-9007(98)00171-3. PMID 9990575
- [Background] Detsky AS, McLaughlin JR, Baker JP, Johnston N, Whittaker S, Mendelson RA, Jeejeebhoy KN. What is subjective global assessment of nutritional status? JPEN J Parenter Enteral Nutr. 1987 Jan-Feb;11(1):8-13. doi: 10.1177/014860718701100108. PMID 3820522
- [Background] Alwall N. Historical perspective on the development of the artificial kidney. Artif Organs. 1986 Apr;10(2):86-99. doi: 10.1111/j.1525-1594.1986.tb02526.x. No abstract available. PMID 3521553
- [Background] Correa-Rodriguez M, Pocovi-Gerardino G, Callejas-Rubio JL, Fernandez RR, Martin-Amada M, Cruz-Caparros MG, Ortego-Centeno N, Rueda-Medina B. The Prognostic Nutritional Index and Nutritional Risk Index Are Associated with Disease Activity in Patients with Systemic Lupus Erythematosus. Nutrients. 2019 Mar 16;11(3):638. doi: 10.3390/nu11030638. PMID 30884776
- [Background] Aparicio-Soto M, Sanchez-Hidalgo M, Alarcon-de-la-Lastra C. An update on diet and nutritional factors in systemic lupus erythematosus management. Nutr Res Rev. 2017 Jun;30(1):118-137. doi: 10.1017/S0954422417000026. Epub 2017 Mar 15. PMID 28294088
- [Background] Allanore Y, Simms R, Distler O, Trojanowska M, Pope J, Denton CP, Varga J. Systemic sclerosis. Nat Rev Dis Primers. 2015 Apr 23;1:15002. doi: 10.1038/nrdp.2015.2. PMID 27189141